CLINICAL TRIAL: NCT07128498
Title: Tinkering to Flex Ur Brain (Tinker-FUN): A Cognitive Flexibility Pilot Program for Community Dwelling Older Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 202500918
Record Dates: First submitted 2025-08-13; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Cognition Improvement
Keywords: Older Adults; Cognition; Cognitive Flexibility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tinker-FUN (Experimental): Intervention arm utilizing the Tinker-FUN program
  Interventions: Behavioral: Tinker-Fun

INTERVENTIONS:
Behavioral: Tinker-Fun — A cognitive flexibility intervention revolves around a hands-on experience where participants design and build a craft or device. The process emphasizes active learning through observing, exploring, t

SUMMARY:
The Tinker-FUN program is a cognitive flexibility intervention designed to help older adults adapt to aging and live independently. While cognitive training is an effective way to mitigate cognitive decline, current methods do not focus on cognitive flexibility, an essential aspect of managing daily activities as one ages. The intervention aims to address this gap by offering engaging tinkering activities designed for older adults. Before expanding to a larger clinical trial, the current proposal seeks to test its feasibility among community-dwelling older adults in US.

ELIGIBILITY:
Inclusion Criteria:

* Mini MoCA Score >12

Exclusion Criteria:

* Diagnosed or self-reported cognitive impairment
* Diagnosed or self-reported psychiatric disorders
* Diagnosed or self-reported neurological disorders

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
NIH Toolbox Cognition Battery Composite Score | From Baseline to the end of the intervention 3 months later.
  This score represents an overall measure of cognitive ability and is derived from the cognitive measures from the NIH Toolbox.

SECONDARY OUTCOMES:
Task Switching Paradigm Score | Baseline to the end of the 3 month intervention.
  The Task Switching Paradigm measures cognitive flexibility.

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Te Wu, PhD, Principal Investigator — University of Florida

IPD SHARING:
Plan to Share IPD: No
IPD will not be included in the data sets which will be analyzed for this study. Published data will comprise of summery scores and other statistical elements not individual level data.